CLINICAL TRIAL: NCT07281209
Title: A Single-Arm Phase II Clinical Study of SHR-A1811 Combined With Adebelimumab as Neoadjuvant Therapy for Resectable HER2-Altered Non-Small Cell Lung Cancer
Brief Title: A Study of SHR-A1811 Combined With Adebelimumab as Neoadjuvant Therapy for Resectable HER2-Altered Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Ziming Li, Chief Physician, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IS25205
Record Dates: First submitted 2025-11-19; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: NSCLC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A1811 combined with Adebelimumab (Experimental)
  Interventions: Drug: SHR-A1811 + Adebrelimab

INTERVENTIONS:
Drug: SHR-A1811 + Adebrelimab — This study evaluates a novel, chemotherapy-free neoadjuvant regimen uniquely combining the HER2-targeting ADC SHR-A1811 with the anti-PD-L1 antibody Adebrelimab. This specific combination of a HER2-ADC and an immune checkpoint inhibitor in the pre-operative setting for HER2-altered NSCLC is the primary feature distinguishing this intervention.

SUMMARY:
This is a prospective, single-arm, multi-center Phase II clinical trial designed to evaluate the efficacy and safety of neoadjuvant therapy with SHR-A1811 in combination with Adebelimumab in patients with resectable, early-stage non-small cell lung cancer (NSCLC) harboring HER2 alterations.

ELIGIBILITY:
Inclusion Criteria:

1. Having sufficient understanding of this study and being willing to sign the informed consent form (ICF);
2. Aged 18-75 years, male or female;
3. Treatment-naive, histologically confirmed resectable, stage II, IIIA, IIIB (AJCC staging system, version 9) NSCLC
4. HER2 alterations identified by histological specimens;
5. Measurable lesions based on the response evaluation criteria in solid tumors version 1.1 (RECIST v1.1);
6. ECOG score 0-1;
7. No contraindications to immunotherapy;
8. Adequate organ function:
9. Being willing and able to comply with the visits, treatment plan, laboratory examinations and other study procedures scheduled in the study;
10. Pulmonary function being able to withstand the planned surgery evaluated by surgeons;
11. Women of childbearing potential must undergo a serum pregnancy test within 1 week prior to the first dose and the result must be negative. Female patients of childbearing potential and male subjects whose partners are women of childbearing potential must agree to use highly effective contraceptive methods during the study period and within 180 days after the last dose of study drug

Exclusion Criteria:

1. Known EGFR sensitizing mutations or ALK fusions.
2. Malignant pleural effusion. Drainable effusions during screening require thoracentesis to rule out malignancy.
3. Prior anticancer therapy (radiotherapy, chemotherapy, immunotherapy), except curatively treated NSCLC with ≥5 years recurrence-free. Anticancer Chinese herbal medicine is allowed if stopped ≥2 weeks prior.
4. Active or history of autoimmune diseases (e.g., uveitis, hepatitis, vasculitis, thyroiditis). Exceptions include: resolved childhood asthma, vitiligo, psoriasis, or alopecia without systemic treatment. Patients requiring bronchodilators are excluded.
5. Immunodeficiency (e.g., HIV), active Hepatitis B (HBsAg+ & HBV DNA ≥500 IU/mL), or active Hepatitis C (HCV Ab+ & detectable HCV RNA). Resolved HBV infection (anti-HBc+, HBsAg-) is allowed.
6. Uncontrolled third-space fluid accumulation requiring repeated drainage.
7. Significant proteinuria (urine protein ≥++ and 24-hour protein ≥1.0 g) or severe hepatic/renal impairment.
8. Systemic corticosteroids (>10 mg/day prednisone equivalent) or immunosuppressants within 14 days prior to first dose. Inhaled/topical steroids or physiologic replacement doses are permitted.
9. Antitumor vaccines or immunostimulatory agents within 1 month prior to first dose.
10. Systemic immunosuppressive therapy within 2 weeks prior to first dose or anticipated need during the study. Short-term, low-dose use may be permitted after Medical Monitor approval.
11. Concurrent participation in another interventional clinical trial or prior interventional drug within 4 weeks (or 5 half-lives). Non-interventional study participation is allowed.
12. Known or suspected interstitial lung disease, or other significant pulmonary conditions that may interfere with drug-related pulmonary toxicity evaluation.
13. Severe cardiovascular disease, including: clinically significant arrhythmias; QTc ≥450 ms (male) or ≥470 ms (female); NYHA Class ≥III heart failure; or LVEF <50%.
14. Severe infection within 4 weeks prior to first dose, or active infection requiring therapeutic antibiotics within 2 weeks prior (prophylactic antibiotics allowed).
15. Active tuberculosis within 1 year prior to first dose.
16. Major surgery within 28 days prior to first dose.
17. History of allogeneic organ or stem cell transplantation.
18. Pregnancy, lactation, or unwillingness to use effective contraception.
19. Known allergy or hypersensitivity to SHR-A1811/Adebelimumab or their excipients.
20. History of psychoactive drug abuse, alcohol abuse, or drug addiction. 21 Any other condition that may compromise patient safety or study compliance, per investigator's judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
pCR rate | up to 7 weeks after neoadjuvant
  Pathological Complete Response (pCR) Rate is defined as the percentage of participants having an absence of residual invasive cancer in resected lung specimens and lymph nodes following completion of neoadjuvant therapy.

SECONDARY OUTCOMES:
MPR rate | up to 7 weeks after neoadjuvant
  Major Pathological Response (MPR) Rate is defined as the percentage of participants having ≤10% viable tumor cells in the resected primary tumor and all resected lymph nodes in neoadjuvant therapy.
ORR | up to 7 weeks after neoadjuvant
  Objective Response Rate (ORR) is defined as the percentage of participants achieving complete response (CR) and partial response (PR) for tumor volume reduction and maintaining the minimum duration requirement based on RECIST v1.1
EFS | up to 3 years
  Event Free Survival (EFS) is defined as the time from randomization until radiographic disease progression, local progression precluding surgery, inability to resect the tumor, local or distant recurrence, or death due to any cause.
OS | up to 3 years
  Overall survival (OS) is defined as the time from randomization until death from any cause.
Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) | 90 days after the last administration
  Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0